CLINICAL TRIAL: NCT05548920
Title: Preoperative Ultrasound Guided Evaluation of Subclavian Vein Collapsibility Index and Inferior Vena Cava Collapsibility Index as Predictors of Hypotension After Induction of General Anesthesia in Major Onco-surgery
Brief Title: Preoperative Ultrasound Guided Evaluation of SVC-CI and IVC -CI as Predictors of Hypotension After Induction of Anaesthesia in Major Onco-surgery
Acronym: SVC IVC CI
Status: Completed | Type: Observational
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Senior Consultant, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: SCV IVC Collapsibility
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Total Fluid Volume Decreased

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasound guided Superior Vena Cava Collapsibility Index (SVC - CI): Preoperative ultrasound guided Superior Vena Cava collapsibility Index will be measured with patient breathing spontaneously and on deep inspiration.
  Interventions: Other: Ultrasound guided Superior Vena Cava Collapsibility Index
- Ultrasound Guided Inferior Vena Cava Collapsibility Index (IVC -CI): Preoperative Ultrasound guided Inferior Vena Cava collapsibility Index will be measured with patient breathing spontaneously and on deep inspiration.
  Interventions: Other: Inferior Vena Cava Collapsibility Index

INTERVENTIONS:
Other: Ultrasound guided Superior Vena Cava Collapsibility Index — Preoperative Ultrasound guided Superior Vena Cava Collapsibility Index will be measured
  Groups: Ultrasound guided Superior Vena Cava Collapsibility Index (SVC - CI)
Other: Inferior Vena Cava Collapsibility Index — Preoperative Inferior Vena Cava Collapsibility Index will be measured.
  Groups: Ultrasound Guided Inferior Vena Cava Collapsibility Index (IVC -CI)

SUMMARY:
Patients undergoing major Oncosurgeries are fluid deficit due to preoperative fasting , inadequate intake due to disease hence prone to development of hypotension after induction of general anaesthesia owing to vasodilatory effects of anesthetic induction agents. Investigators plan study to measure ultrasound guided Superior Vena Cava and Inferior Vena Cava collapsibility Index as predictors of hypotension after induction of General anaesthesia.

DETAILED DESCRIPTION:
Investigators plan prospective study , written informed will be taken from all included patients. In the OR 5 lead ECG, NIBP,SPO2 monitors will be attached , patients will be explained about Ultrasound imaging . Preinduction using SONOSITE EDGE II ultrasonography machine and placing high frequency linear array probe (6-13 Hz) beneath the middle of the clavicle aligned in deltopectoral groove to obtain short axis view of Subclavian/Infraclavicular axillary vein in B-Mode (2-D imaging). Doppler pulse waveform and minimum and maximum diameter measurements of SVC will be obtained in M-mode , both during spontaneous breathing and after deep inspiration, using digital calipers after freezing the image. The collapsibility index CI will be calculated using the following equation SCV AV CI = (dSCV max- dSCV min)/ dSCV max ×100.

A phased array or cardiac ultrasound probe (1-5Hz) will be placed in the subxiphoid window to view IVC at the junction of IVC with right atrium .Then the transducer will be adjusted to obtain the long axis view of IVC. Doppler pulse waveform will be obtained to ensure imaging of IVC and then in the M mode the minimum and maximum diameter measurements of IVC will be obtained both during spontaneous breathing and after deep inspiration, using digital calipers after freezing the image. The collapsibility index CI will calculated using the following equation:IVC CI = (dIVCmax- dIVCmin )/ dIVCmax ×100 . In all the patients both SVC and IVC -CI will be calculated.

All patients will receive standard General Anesthesia with IV Fentanyl 1-2 mcg/kg , Sleeping dose propofol , Atracurium 0.5mg/kg and orally placed Endotracheal tube.The heart rate (HR) and mean arterial pressure (MAP) will be recorded in two phases .Intraoperative hypotension (IOH) been defined as MAP<60mmHg or >30%decrease in MAP from baseline.

1. Post induction phase: Readings will be taken at 1 min intervals from the start of induction till intubation (upto 5 minutes) and
2. Post intubation phase: Readings will be taken at 2 min intervals upto 10 min and at 5 min intervals up to 30 mins or till incision . Each hypotensive episode encountered will be treated with leg lifting first (lifting both lower extremities for 2 minutes by technical staff) , if hypotension persists then IV Ephedrine 6 mg boluses will be given . All patients will receive preloading 200ml crystalloids prior to induction of anesthesia .

ELIGIBILITY:
Inclusion Criteria:

* Patients belonging to ASA Grade I,II,III
* For major Oncosurgery under general anaesthesia

Exclusion Criteria:

* Patient refusal
* BMI>30
* Emergency surgery
* Preoperative Hypotension MAP < 70 mmHg
* LVEF<40%
* Difficult Airway
* Nasal Intubation
* Inability to obtain good ultrasound images of SCV and IVC .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing major Onco-surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
To compare Subclavian Vein Collapsibility Index in percentage with Inferior Vena Cava Collapsibility Index in percentage as predictor of hypotension after induction of General anaesthesia | 30 minutes prior to induction of anaesthesia
  Preoperative Ultrasound guided Subclavian / Infraclavicular Axillary Vein Collapsibility Index and Inferior Vena Cava Collapsibility Index was measured with spontaneous breathing and on deep inspiration.

SECONDARY OUTCOMES:
To evaluate the sensitivity of SVC -CI and IVC -CI as a predictor of hypotension after induction of General anesthesia . | 30 minutes prior to induction of anaesthesia
  Preoperative US Guided SVC-CI in percentage and IVC -CI in percentage values will be obtained and statistical analysis will be done

CONTACTS AND LOCATIONS:
Overall Officials: Anita C Kulkarni, MD, Principal Investigator — Senior Consultant
Locations (1):
- Rajiv Gandhi Cancer Institute and Research Centre, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choi MH, Chae JS, Lee HJ, Woo JH. Pre-anaesthesia ultrasonography of the subclavian/infraclavicular axillary vein for predicting hypotension after inducing general anaesthesia: A prospective observational study. Eur J Anaesthesiol. 2020 Jun;37(6):474-481. doi: 10.1097/EJA.0000000000001192. PMID 32205573
- [Result] Kaptein YE, Kaptein EM. Comparison of subclavian vein to inferior vena cava collapsibility by ultrasound in acute heart failure: A pilot study. Clin Cardiol. 2022 Jan;45(1):51-59. doi: 10.1002/clc.23758. Epub 2021 Dec 21. PMID 34931333